CLINICAL TRIAL: NCT04202471
Title: Preoperative Chlorhexidine Cloths to Reduce Surgical Site Infection in Non-Scheduled Cesarean Deliveries
Brief Title: Chlorhexidine Cloths to Reduce Surgical Site Infection in Cesarean Deliveries
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Moti Gulersen, Principal Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19-1040
Record Dates: First submitted 2019-12-14; First posted 2019-12-17 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Surgical Site Infection
Keywords: Chlorhexidine Cloth; Surgical Site Infection; Non-scheduled cesarean delivery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Chlorhexidine Cloth (Experimental): The intervention group will be women undergoing non-scheduled cesarean delivery randomized to receive preoperative abdominal application of 2% chlorhexidine cloths.
  Interventions: Device: Chlorhexidine Cloth
- Standard Preoperative Care (No Intervention): The no intervention group will be women undergoing non-scheduled cesarean delivery randomized to receive standard preoperative care.

INTERVENTIONS:
Device: Chlorhexidine Cloth — 2% chlorhexidine gluconate cloth
  Arms: Chlorhexidine Cloth

SUMMARY:
Pregnancy-associated infection represents a major cause of maternal morbidity and mortality. Cesarean delivery is the most common major surgical procedure and is associated with a rate of surgical site infection (SSI) that is approximately 5-10 times the rate for vaginal delivery. Efforts to reduce the risk of SSIs in this patient population include the use of preoperative antibiotic prophylaxis in addition to skin and vaginal antiseptic preparations.Nevertheless, the rate of SSI in women undergoing non-scheduled cesarean delivery is up to 18%, a significant number that contributes to prolonged hospital stays and increased health care costs.

Every effort should be made to reduce this major cause of pregnancy-associated morbidity and mortality to aid in the care of patients and reduce the associated prolonged hospital stays, readmission rates and health care costs. Studies have shown that preoperative application of chlorhexidine cloths reduces the risk of SSI, however this is based on literature in the orthopedic and intensive care patients. The efficacy of this intervention has not been studied in obstetric patients undergoing cesarean delivery. Furthermore, obstetric patients undergoing non-scheduled cesarean delivery represent a target population as it is thought that infectious morbidity is higher in this patient population. Therefore, there is a need for this trial to determine if this intervention is effective in reducing the rate of postoperative SSIs.

DETAILED DESCRIPTION:
This randomized clinical trial will be investigating the use of preoperative chlorhexidine cloths, a chemical skin antiseptic agent effective on gram positive and gram negative bacteria, as an intervention to reduce the rate of surgical site infections (SSIs). The intervention group will be women undergoing non-scheduled cesarean delivery randomized to receive preoperative abdominal application of 2% chlorhexidine cloths. The control group will be women undergoing non-scheduled cesarean delivery randomized to receive standard preoperative care. The impact on women's health is significant, as a reduction in SSIs in this prevalent patient population can reduce the number of prolonged hospital stays, outpatient follow-ups for infection, hospital readmissions and health care costs.

ELIGIBILITY:
Inclusion Criteria:

* undergoing non-scheduled cesarean delivery > 23 weeks gestation

Exclusion Criteria:

* allergy to chlorhexidine, emergency cesarean delivery, evidence of infection at operative site

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of surgical site infection | Up to 6 weeks after cesarean delivery

SECONDARY OUTCOMES:
Hospital length of stay | Up to 6 weeks after cesarean delivery
Number of office visits | Up to 6 weeks after cesarean delivery
Number of hospital readmissions for infection-related complications | Up to 6 weeks after cesarean delivery
Rate of endometritis | Up to 6 weeks after cesarean delivery
Rate of positive wound culture from wound | Up to 6 weeks after cesarean delivery

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

REFERENCES:
- [Background] Carter EB, Temming LA, Fowler S, Eppes C, Gross G, Srinivas SK, Macones GA, Colditz GA, Tuuli MG. Evidence-Based Bundles and Cesarean Delivery Surgical Site Infections: A Systematic Review and Meta-analysis. Obstet Gynecol. 2017 Oct;130(4):735-746. doi: 10.1097/AOG.0000000000002249. PMID 28885421
- [Background] Shree R, Park SY, Beigi RH, Dunn SL, Krans EE. Surgical Site Infection following Cesarean Delivery: Patient, Provider, and Procedure-Specific Risk Factors. Am J Perinatol. 2016 Jan;33(2):157-64. doi: 10.1055/s-0035-1563548. Epub 2015 Sep 7. PMID 26344010
- [Background] Moulton LJ, Munoz JL, Lachiewicz M, Liu X, Goje O. Surgical site infection after cesarean delivery: incidence and risk factors at a US academic institution. J Matern Fetal Neonatal Med. 2018 Jul;31(14):1873-1880. doi: 10.1080/14767058.2017.1330882. Epub 2017 Jun 8. PMID 28502188
- [Background] Tuuli MG, Liu J, Stout MJ, Martin S, Cahill AG, Odibo AO, Colditz GA, Macones GA. A Randomized Trial Comparing Skin Antiseptic Agents at Cesarean Delivery. N Engl J Med. 2016 Feb 18;374(7):647-55. doi: 10.1056/NEJMoa1511048. Epub 2016 Feb 4. PMID 26844840
- [Background] Springel EH, Wang XY, Sarfoh VM, Stetzer BP, Weight SA, Mercer BM. A randomized open-label controlled trial of chlorhexidine-alcohol vs povidone-iodine for cesarean antisepsis: the CAPICA trial. Am J Obstet Gynecol. 2017 Oct;217(4):463.e1-463.e8. doi: 10.1016/j.ajog.2017.05.060. Epub 2017 Jun 7. PMID 28599898
- [Background] Boyce JM. Best products for skin antisepsis. Am J Infect Control. 2019 Jun;47S:A17-A22. doi: 10.1016/j.ajic.2019.03.012. PMID 31146845
- [Background] Ahmed MR, Aref NK, Sayed Ahmed WA, Arain FR. Chlorhexidine vaginal wipes prior to elective cesarean section: does it reduce infectious morbidity? A randomized trial. J Matern Fetal Neonatal Med. 2017 Jun;30(12):1484-1487. doi: 10.1080/14767058.2016.1219996. Epub 2016 Sep 1. PMID 27583685
- [Background] Connery SA, Yankowitz J, Odibo L, Raitano O, Nikolic-Dorschel D, Louis JM. Effect of using silver nylon dressings to prevent superficial surgical site infection after cesarean delivery: a randomized clinical trial. Am J Obstet Gynecol. 2019 Jul;221(1):57.e1-57.e7. doi: 10.1016/j.ajog.2019.02.053. Epub 2019 Mar 5. PMID 30849351
- [Background] Kapadia BH, Elmallah RK, Mont MA. A Randomized, Clinical Trial of Preadmission Chlorhexidine Skin Preparation for Lower Extremity Total Joint Arthroplasty. J Arthroplasty. 2016 Dec;31(12):2856-2861. doi: 10.1016/j.arth.2016.05.043. Epub 2016 May 31. PMID 27365294
- [Background] Zywiel MG, Daley JA, Delanois RE, Naziri Q, Johnson AJ, Mont MA. Advance pre-operative chlorhexidine reduces the incidence of surgical site infections in knee arthroplasty. Int Orthop. 2011 Jul;35(7):1001-6. doi: 10.1007/s00264-010-1078-5. Epub 2010 Jun 20. PMID 20563806
- [Background] Kapadia BH, Johnson AJ, Daley JA, Issa K, Mont MA. Pre-admission cutaneous chlorhexidine preparation reduces surgical site infections in total hip arthroplasty. J Arthroplasty. 2013 Mar;28(3):490-3. doi: 10.1016/j.arth.2012.07.015. Epub 2012 Oct 29. PMID 23114192
- [Background] Dixon JM, Carver RL. Daily chlorohexidine gluconate bathing with impregnated cloths results in statistically significant reduction in central line-associated bloodstream infections. Am J Infect Control. 2010 Dec;38(10):817-21. doi: 10.1016/j.ajic.2010.06.005. PMID 21093698
- [Background] Popovich KJ, Hota B, Hayes R, Weinstein RA, Hayden MK. Effectiveness of routine patient cleansing with chlorhexidine gluconate for infection prevention in the medical intensive care unit. Infect Control Hosp Epidemiol. 2009 Oct;30(10):959-63. doi: 10.1086/605925. PMID 19712033
- [Background] Kuyyakanond T, Quesnel LB. The mechanism of action of chlorhexidine. FEMS Microbiol Lett. 1992 Dec 15;100(1-3):211-5. doi: 10.1111/j.1574-6968.1992.tb14042.x. PMID 1335944
- [Background] Darouiche RO, Wall MJ Jr, Itani KM, Otterson MF, Webb AL, Carrick MM, Miller HJ, Awad SS, Crosby CT, Mosier MC, Alsharif A, Berger DH. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. N Engl J Med. 2010 Jan 7;362(1):18-26. doi: 10.1056/NEJMoa0810988. PMID 20054046
- [Background] DeBaun B. Evaluation of the antimicrobial properties of an alcohol-free 2% chlorhexidine gluconate solution. AORN J. 2008 May;87(5):925-33. doi: 10.1016/j.aorn.2008.02.001. PMID 18489920
- [Background] Edmiston CE Jr, Krepel CJ, Seabrook GR, Lewis BD, Brown KR, Towne JB. Preoperative shower revisited: can high topical antiseptic levels be achieved on the skin surface before surgical admission? J Am Coll Surg. 2008 Aug;207(2):233-9. doi: 10.1016/j.jamcollsurg.2007.12.054. Epub 2008 May 23. PMID 18656052
- [Background] Edmiston CE Jr, Seabrook GR, Johnson CP, Paulson DS, Beausoleil CM. Comparative of a new and innovative 2% chlorhexidine gluconate-impregnated cloth with 4% chlorhexidine gluconate as topical antiseptic for preparation of the skin prior to surgery. Am J Infect Control. 2007 Mar;35(2):89-96. doi: 10.1016/j.ajic.2006.06.012. PMID 17327187